CLINICAL TRIAL: NCT02994433
Title: NMDA Receptor Antagonist Nitrous Oxide Targets Affective Brain Circuits
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: remaining visits and enrollment terminated due to the pandemic
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 201606120
Record Dates: First submitted 2016-12-02; First posted 2016-12-15 (Estimated); Last update posted 2021-08-02 (Actual); Status verified 2021-07

CONDITIONS: Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nitrous Oxide (Experimental): One hour inhalation of nitrous oxide
  Interventions: Drug: Nitrous Oxide; Device: MRI
- Placebo Gas (Placebo Comparator): One hour inhalation of placebo gas
  Interventions: Drug: Placebo gas; Device: MRI

INTERVENTIONS:
Drug: Nitrous Oxide — Nitrous oxide, an odorless, colorless gas typically used as an induction agent for general anesthesia or for dental sedation, is a known N-methyl-D-aspartate (NMDA) antagonist. It will be given at 50% nitrous oxide/50% oxygen in this study.
  Other Names: laughing gas
  Arms: Nitrous Oxide
Drug: Placebo gas — Placebo gas given at 50% nitrogen [inert]/50% oxygen.
  Arms: Placebo Gas
Device: MRI — MRIs done on all participants, this is a tool we are using to measure outcomes. No treatment is from an MRI.

SUMMARY:
Most clinical major depression responds to standard treatments (medication and psychotherapy); however, a significant subset of depressed patients (15-20%) do not respond to these treatments and are referred to as treatment-resistant major depression (TRMD). New treatments for TRMD are needed, and one promising line of research are drugs known as N-methyl-D-aspartate (NMDA) glutamate receptor antagonists. In a recent pilot study, our group demonstrated that the NMDA antagonist nitrous oxide is effective in TRMD. This application proposes to take the next important step in understanding how nitrous oxide exerts its effects in the human brain by using state-of-the-art brain neuroimaging (functional connectivity magnetic resonance imaging) in a group of non-depressed, healthy volunteers and comparing the results to a group of TRMD patients.

This study involves exposing 20 non-depressed healthy participants and 20 TRMD participants to nitrous oxide and a placebo gas, to compare their brain images before and after each of the inhalation sessions. Sessions will be separated by at least one month to prevent treatment effects from carrying over into the following session. All willing and eligible subjects will undergo up to six functional connectivity MRI scans, and two inhalation sessions. Functional imaging in the brain will allow us to trace the interconnections between various parts of the brain, including those involved with emotion and depression.

Other procedures will involve screening materials to ensure safety of the participants before beginning the study (i.e. no MRI scan contraindications) and that subjects meet eligibility criteria to being in the targeted age range, depression/non-depressed state, neurological disorder history, and no medication exclusions.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* Right-handed
* Controls: Not meet The Fourth Edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) criteria for major depressive disorder (MDD) by scoring ≤7 on the Hamilton Depression Rating Scale (HDRS), 17-item; Treatment-Resistant Major Depression (TRMD) patients: Must meet a ≥17 score on the HDRS.
* Controls: Must not have any history of depression as determined by reported history and medical record review; TRMD: Documented (chart review) failure to respond to ≥3-4 adequate dose/duration antidepressant treatments; ≥1 in the current depressive episode.
* Good command of the English language

Exclusion Criteria:

* Meets criteria for any DSM-IV Axis I diagnosis as documented in medical records and as determined by structured clinical interview (except MDD for the TRMD group)
* Known primary neurological disorders or medical disorders including dementia, stroke, encephalopathy Parkinson's Disease, brain tumors, multiple sclerosis, seizure disorder, severe cardiac or pulmonary disease
* Any central nervous system active medication as determined by study investigator
* Any known disease affecting drug metabolism and excretion (e.g. renal or liver disease) as determined by study investigator
* Left-handedness
* Not eligible for MRI scans (e.g. history of claustrophobia/implanted metal as per MRI Screening Tool)
* Current use of psychotropic medications, antidepressants, or prescription or non-prescription drugs/herbals intended to treat depression or anxiety (control group only)
* Any recent (within past 12 months) history of substance dependence or abuse, determined by reported history or urine drug screen
* Ability to become pregnant and not using effective contraception
* Contraindication against the use of nitrous oxide:

  1. Pneumothorax
  2. Bowel obstruction
  3. Middle ear occlusion
  4. Elevated intracranial pressure
  5. Chronic cobalamin and/or folate deficiency treated with folic acid or vitamin B12
  6. Pregnant patients
  7. Breastfeeding women
* Inability to provide informed consent
* Any other factor that in the investigators' judgment may affect patient safety or compliance (e.g. distance greater than 100 miles from clinic).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2017-01-27 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Comparison of functional connectivity between default mode network of treatment-resistant depressed and non-depressed participants | 2 hours after inhalation
  Functional connectivity is measured between groups after inhaling nitrous oxide/placebo using an individual seed-voxel z map and pared t-test group analysis to identify effects on inter-regional connectivity.
Comparison of functional connectivity between affective network of treatment-resistant depressed and non-depressed participants | 2 hours after inhalation
  Functional connectivity is measured between groups after inhaling nitrous oxide/placebo using an individual seed-voxel z map and pared t-test group analysis to identify effects on inter-regional connectivity.
Comparison of functional connectivity between cognitive control network of treatment-resistant depressed and non-depressed participants | 2 hours after inhalation
  Functional connectivity is measured between groups after inhaling nitrous oxide/placebo using an individual seed-voxel z map and pared t-test group analysis to identify effects on inter-regional connectivity.
Comparison of functional connectivity between dorsal nexus of treatment-resistant depressed and non-depressed participants | 2 hours after inhalation
  Functional connectivity is measured between groups after inhaling nitrous oxide/placebo using an individual seed-voxel z map and pared t-test group analysis to identify effects on inter-regional connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Charles R Conway, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Conway CR, Palanca BJA, Zeffiro T, Gott BM, Brown F, de Leon V, Barnes L, Nguyen T, Xiong W, Lessov-Schlaggar CN, Espejo G, Mennerick S, Zorumski CF, Nagele P. Nitrous Oxide Alters Functional Connectivity in Medial Limbic Structures in Treatment-Resistant Major Depression. medRxiv [Preprint]. 2024 Aug 17:2024.08.12.24311729. doi: 10.1101/2024.08.12.24311729. PMID 39185528
- [Derived] de Leon VC, Kumar A, Nagele P, Palanca BJ, Gott B, Janski A, Zorumski CF, Conway CR. Nitrous Oxide Reduced Suicidal Ideation in Treatment-Resistant Major Depression in Exploratory Analysis. J Clin Psychiatry. 2023 Aug 16;84(5):22br14725. doi: 10.4088/JCP.22br14725. No abstract available. PMID 37585253